CLINICAL TRIAL: NCT01353378
Title: Use of Dexmedetomidine in Children Undergoing Oral Maxillofacial Surgery to Decrease Emergence Delirium
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was not approved by Hospital's Medical Ethics Committee.
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Rong Hu, attending in anesthesiology department, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: JYMZK-001
Record Dates: First submitted 2011-04-21; First posted 2011-05-13 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Delirium
Keywords: dexmedetomidine; emergence delirium; sevoflurane anesthesia; preschool children; oral maxillofacial surgery
MeSH Terms: conditions — Delirium; Emergence Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dexmedetomidine (Experimental): intravenously injecting 0.125microgram/kg and 0.25microgram/kg within 10 minutes as soon as the operation begins respectively.
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine — Intravenously injecting 0.125microgram/kg for 10ml IV(in the vein)in group 1, 0.25microgram/kg for 10ml in group 2 within 10 minutes as soon as the operation begin. The control group receives 10mlsaline in 10 minutes.
  Other Names: dexmedetomidine hydrochloride injection

SUMMARY:
The purpose of this study is to determine whether dexmedetomidine is effective in the treatment of emergence delirium of preschool children undergoing oral maxillofacial surgery.

DETAILED DESCRIPTION:
Emergence delirium is a common side effect of sevoflurane anesthesia in children. Dexmedetomidine, because of its sedative and analgesic properties, might be useful for the management of this adverse effect. In the pediatric population, it has been shown to provide sedation for magnetic resonance imaging. Intravenously, it is has been shown to decrease emergence delirium following sevoflurane based anesthesia. The ability to administer a medication intravenously might solve the problem of emergence delirium and emergence agitation posed by the young patients undergoing oral maxillofacial surgery.

ELIGIBILITY:
Inclusion Criteria:

* preschool children undergoing oral maxillofacial surgery

Exclusion Criteria:

* mental diseases
* history of neural system disease
* sedative medication history
* anticipated difficult airway

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
post anesthesia emergence delirium scale(PAED scale) | 2 hours post-surgery
  evaluate children's PAED scale score 2 hours post-surgery

SECONDARY OUTCOMES:
Children's Hospital of Eastern Ontario Pain Scale(CHEOP scale) | 2 hours post-surgery
  evaluate children's CHEOP scale score 2 hours post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jiang, MD, PHD, Study Director — Department of Anesthesiology, Shanghai Ninth People's Hospital affiliated to Shanghai Jiao Tong University, School of Medicine; Rong Hu, MD, Principal Investigator — Department of Anesthesiology, Shanghai Ninth People's Hospital affiliated to Shanghai Jiao Tong University, School of Medicine
Locations (1):
- Shanghai Ninth People's Hospital affiliated to Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality, China